CLINICAL TRIAL: NCT03006354
Title: Nasal High Frequency Oscillatory Ventilation Versus Nasal Continuous Positive Airway Pressure in Late-Preterm and Term Infants With Transient Tachypnea of the Newborn: a Randomized Controlled Trial
Brief Title: nHFOV Versus nCPAP in Transient Tachypnea of the Newborn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Mehmet Cizmeci, Associate Professor of Pediatrics, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-KAEK-25 2016/22-06
Record Dates: First submitted 2016-12-28; First posted 2016-12-30 (Estimated); Last update posted 2023-12-06 (Actual); Status verified 2017-03

CONDITIONS: Transient Tachypnea of the Newborn
Keywords: high frequency oscillatory ventilation; newborn; noninvasive ventilation; transient tachypnea of the newborn
MeSH Terms: conditions — Transient Tachypnea of the Newborn | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nHFOV (Experimental): Ventilator-derived nHFOV will be administered using binasal prongs. Standard Device: Leoni-Plus or Leoni-2 Ventilator, Heinen Löwenstein, Germany Initial nHFOV settings are: MAP: 8cmH2O, Frequency:10 MHz, Amplitude:35 cmH2O (will be adjusted to achieve adequate chest wall vibration), I:E=1:1 and FiO2: adjusted to keep preductal sPO2 between %90-95.
  Failure is defined as FiO2 requirement of >%60, capillary blood gas obtained at the 4th hour of therapy showing pH<7.20 or pCO2>65 cmH2O.
  When nHFOV failure occurs, nasal intermittent positive pressure ventilation (nIPPV) will be applied as a rescue therapy with the following settings: Frequency:30/min, PIP:18 cmH2O, PEEP:6 cmH2O, inspiration time:0.50 sec., inspiratory flow:10 L/min, FiO2:adjusted to keep preductal sPO2 between %90-95.
  Interventions: Device: nHFOV
- nCPAP (Active Comparator): Ventilator-derived nCPAP will be administered using binasal prongs. Standard Device: Leoni-Plus or Leoni-2 Ventilator, Heinen Löwenstein, Germany Initial nCPAP settings are: PEEP:6 cmH2O and FiO2: adjusted to keep preductal sPO2 between %90-95.
  Failure is defined as FiO2 requirement of >%60, capillary blood gas obtained at the 4th hour of therapy showing pH<7.20 or pCO2>65 cmH2O.
  When nCPAP failure occurs, nasal intermittent positive pressure ventilation (nIPPV) will be applied as a rescue therapy with the following settings: Frequency:30/min, PIP:18 cmH2O, PEEP:6 cmH2O, inspiration time:0.50 sec., inspiratory flow:10 L/min, FiO2:adjusted to keep preductal sPO2 between %90-95.
  Interventions: Device: nCPAP

INTERVENTIONS:
Device: nHFOV — Ventilator (Leoni-Plus Ventilator, Heinen-Lowenstein, Germany) derived high frequency oscillatory ventilation, using binasal prongs
  Other Names: nasal high frequency oscillatory ventilation
  Arms: nHFOV
Device: nCPAP — Ventilator (Leoni-Plus or Leoni-2 Ventilator, Heinen-Lowenstein, Germany) derived high frequency oscillatory ventilation, using binasal prongs
  Other Names: nasal continuous positive airway pressure
  Arms: nCPAP

SUMMARY:
In this prospective, randomised clinical trial the investigators aim to assess if nasal high frequency oscillatory ventilation (nHFOV) could be used as the primary modality of respiratory support in late preterm and term infants with transient tachypnea of the newborn requiring non-invasive ventilation.

DETAILED DESCRIPTION:
BACKGROUND: Non-invasive High Frequency Oscillatory Ventilation (nHFOV), aims to combine the efficacy of high frequency ventilation with the gentleness of non-invasive support and current evidence suggests that nHFOV may be superior to other non-invasive modes in terms of supporting alveolar ventilation. There are now several published neonatal studies of nHFOV therapy as a rescue mode even in the premature infants; however to date no studies have been published on the efficacy of nHFOV as a primary mode of non-invasive support. The investigators aim to assess the efficacy of nHFOV in late-preterm and term infants with transient tachypnea of the newborn as the primary mode of non-invasive support.

METHOD: The investigators propose to test the effectiveness of nHFOV in late-preterm and term neonates with transient tachypnea of the newborn (TTN) with a Silverman Score of 4 or above on admission who require non-invasive respiratory support. Nasal high frequency oscillatory ventilation may be effective in decreasing duration of non-invasive respiratory support and total oxygen therapy (H1 hypotheses).

The current literature estimates the incidence of transient tachypnea of the newborn to be 5.7 per 1000 births. Assuming that a 5% difference of the primary outcome between the groups is significant, when the alpha value is set at 0.05 and power of the study at 80%, 220 infants must be recruited for each arm (nCPAP and nHFOV) under investigation.

Chest X-ray, complete blood count, C-reactive protein and capillary blood gas analysis (as per unit protocol) will be obtained upon admission to the neonatal intensive care unit. A Silverman Score will be obtained for each participant upon admission and those with a score of 4 and above will be supported with one of the methods (with randomization).

Initial nHFOV settings are: MAP: 8cmH2O, Frequency:10 MHz, Amplitude:35 cmH2O (will be adjusted to achieve adequate chest wall vibration), I:E=1:1 and FiO2: adjusted to keep preductal sPO2 between %90-95. Initial nCPAP settings are: PEEP:6 cmH2O and FiO2: adjusted to keep preductal sPO2 between %90-95. Failure of the primary mode is defined as FiO2 requirement of >%60, capillary blood gas obtained at the 4th hour of therapy showing pH<7.20 or pCO2>65 cmH2O. When nCPAP or nHFOV failure occurs, nasal intermittent positive pressure ventilation (nIPPV) will be applied as a rescue therapy with the following settings: Frequency:30/min, PIP:18 cmH2O, PEEP:6 cmH2O, inspiration time:0.50 sec., inspiratory flow:10 L/min, FiO2:adjusted to keep preductal sPO2 between %90-95. If the rescue mode fails, the infant will be intubated and conventional mechanical ventilation will be initiated.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age at birth between 34 and 42 weeks of gestation
* Admission to Bursa Yüksek Ihtisas Teaching Hospital, NICU during the first 24 hours of life
* Diagnosis of transient tachypnea of the newborn (TTN) within the first 24 hours of life

Exclusion Criteria:

* Gestational age at birth less than 34 weeks or greater than 42 weeks at birth
* Chest X-ray or lung ultrasound finding indicating another respiratory disorder
* Additional infant diagnosis of major cardiac disease
* Additional infant diagnosis of major pulmonary disease other than TTN
* Additional infant diagnosis of major congenital anomaly with potential to affect respiratory status in the neonatal period
* Additional infant diagnosis of infectious disease process potentially affecting respiratory status in the neonatal period

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Time to cessation of non-invasive positive pressure respiratory support | 72 hours
  Cessation of nasal flaring, grunting and chest wall retractions (Silverman Score of 0) are indicators of readiness for discontinuation non-invasive positive pressure respiratory support.

SECONDARY OUTCOMES:
Time to cessation of supplemental oxygen | 120 hours
  Total duration of oxygen support of >21%
Time to discharge from hospital | 120 hours
  Discharge time

OTHER OUTCOMES:
Pneumothorax | 72 hours
  Number of pneumothoraces requiring tube thoracostomy in each group

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet N Cizmeci, M.D, Study Director — Bursa Yuksek Ihtisas Teaching Hospital
Locations (1):
- University of Health Sciences, Bursa Yuksek Ihtisas Teaching Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fischer HS, Bohlin K, Buhrer C, Schmalisch G, Cremer M, Reiss I, Czernik C. Nasal high-frequency oscillation ventilation in neonates: a survey in five European countries. Eur J Pediatr. 2015 Apr;174(4):465-71. doi: 10.1007/s00431-014-2419-y. Epub 2014 Sep 18. PMID 25227281
- [Result] De Luca D, Dell'Orto V. Non-invasive high-frequency oscillatory ventilation in neonates: review of physiology, biology and clinical data. Arch Dis Child Fetal Neonatal Ed. 2016 Nov;101(6):F565-F570. doi: 10.1136/archdischild-2016-310664. Epub 2016 Jun 28. PMID 27354382
- [Derived] Baldan E, Varal IG, Dogan P, Cizmeci MN. The effect of non-invasive high-frequency oscillatory ventilation on the duration of non-invasive respiratory support in late preterm and term infants with transient tachypnea of the newborn: a randomized controlled trial. Eur J Pediatr. 2023 Oct;182(10):4499-4507. doi: 10.1007/s00431-023-05128-4. Epub 2023 Jul 26. PMID 37491619